CLINICAL TRIAL: NCT06276621
Title: Family Bridge Program Randomized Controlled Trial
Brief Title: Family Bridge Program
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, K. Casey Lion, Principal Investigator, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: STUDY00003564
Record Dates: First submitted 2024-02-05; First posted 2024-02-26 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Healthcare Inequities; General Pediatric Medical Conditions; Healthcare System Navigation; Patient-provider Communication

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Family Bridge Program (Experimental)
  Interventions: Behavioral: Family Bridge Program
- Care as Usual- Resources Only (Active Comparator)
  Interventions: Behavioral: Care as usual - resources only

INTERVENTIONS:
Behavioral: Family Bridge Program — The Family Bridge Program consists of 7 components, delivered by a trained lay navigator, the Guide. The program includes: (1) orientation to the hospital, unit, room, and hospital resources (e.g., toiletries, loaner phone chargers); (2)unmet social needs assessment, followed by connection to appropriate resources (e.g., food vouchers, community-based transportation); (3)communication and cultural preference assessment (eg, preferred language, comfort asking questions, and health-related cultural beliefs), which is communicated to the medical team and documented in the electronic health record;(4)communication coaching for parents/caregivers to help them clarify and practice asking questions of the medical team; (5)emotional support via daily check-ins during the hospital stay; (6)assistance with logistics ; and (7)one follow-up phone call, 2 days post-discharge, to address remaining questions and connect families to ongoing services if needed.
  Arms: Family Bridge Program
Behavioral: Care as usual - resources only — Families randomized to the control arm will receive FBP written resources, which the Guide (and interpreter, as needed) will review with them over ~5-15 minutes one time. This includes information on hospital services (e.g., cafeteria coupons), community resources (e.g., food and housing support), the structure and roles of the medical team, and the daily hospital schedule. Parents will be informed that their child's nurse is available to help them.
  Arms: Care as Usual- Resources Only

SUMMARY:
Pediatric healthcare disparities in the United States (US) remain persistent and pervasive. Suboptimal patient-provider communication plays an important role in creating and maintaining disparate outcomes; this is compounded by mismatches between a family's skills and resources and the complexity of the health system (such as health literacy and system navigation). Few interventions exist to address disparities related to communication and system navigation in the inpatient setting; given the established links between these and disparate clinical outcomes, such interventions are needed. To address this gap, the study team collaborated with parents/caregivers, staff, and providers to develop and pilot-test a novel program to improve navigation ability, communication, and hospital-to-home transition for a diverse population of children and their families, The Family Bridge Program (FBP).

The FBP combines principles of effective patient navigation and communication coaching interventions into a brief and targeted inpatient program. It is designed for a broad population of low-income children, is not disease-specific, is not limited to English proficient families, and is less time-intensive than traditional navigation, to enable provision of support to more families. The FBP, delivered in-person by a trained lay navigator, includes: (1) hospital orientation; (2) unmet social needs screening (e.g., food insecurity); (3) parent communication and cultural preference assessment, relayed to the medical team; (4) communication coaching for parents; (5) emotional support; (6) assistance with care coordination and logistics; and (7) a phone call 2 days post-discharge. Program elements are flexibly delivered based on parent need and interest.

In pilot testing, the program was feasible to deliver, acceptable to parents and providers, and significantly improved parent-reported system navigation ability. The current R01 proposes a two-site randomized controlled trial (RCT) of the effectiveness of FBP among 728 families of low-income children from families who identify as Hispanic, Black, Asian, Native American/Alaska Native, or Pacific Islander. Enrolled families will be randomized 1:1 (stratified by site and language) to FBP or usual care plus written resources. The specific aims of this clinical trial are to (1) Test the effect of the FBP on parent-reported system navigation ability, quality of hospital-to-home transition, diagnosis comprehension, observed communication quality, perceived stress and revisits; (2) Examine whether changes in parent-reported barriers and needs mediate program effects; and (3) Identify subgroups of parents among whom the FBP is more effective. The proposed RCT will use a rigorous design to test a feasible, innovative program to address a critical national problem. If effective, the Family Bridge Program would provide a scalable model for improving health care experiences and outcomes for families of low-income children at risk for disparities, including those who prefer a language other than English for their medical care.

ELIGIBILITY:
Parents/guardians Inclusion Criteria:

* At least 18 years old; there is no maximum age;
* The legal guardian of an eligible child
* Prefer English, Spanish, Somali or Vietnamese for medical care

Children Inclusion Criteria:

* Under 18 years of age at enrollment; there is no minimum age
* Admitted to a general pediatric service at a participating hospital
* Have been admitted within the past 4 days
* Have public or no insurance (as a proxy for low income)
* Have a self- or parent-reported race/ethnicity other than only non-Hispanic white

Parents/guardians Exclusion Criteria:

- None

Children Exclusion Criteria:

* Not already be enrolled in long-term care coordination or patient services navigation
* Not have an admitting diagnosis that is primarily psychiatric (e.g., anorexia nervosa, suicide attempt)
* Not be admitted for suspicion for child abuse.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 728 (Estimated)
Dates: Start 2024-05-07 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
System Navigation Ability | Enrollment and 2-6 weeks after discharge
  Change score -100 to 100, based on 10-item measure of parent self-reported ability to navigate the healthcare system (e.g., ability to schedule appointments or ask questions).
  Each response of Yes (100), Sometimes (50), or No (0) is averaged to create overall score. Change score as difference from enrollment to follow-up
Pediatric Transition Experience Measure (P-TEM) | 2-6 weeks after discharge
  Percent of items with "top-box" score, based on the Pediatric Transition Experience Measure (P-TEM), an 8-item measure to assess hospital-to-home transition. Responses are on Likert scale from 0 to 5, with top-box scoring for overall measure.

SECONDARY OUTCOMES:
Diagnosis Comprehension | 2-6 weeks after discharge
  Discharge diagnosis concordance: 2 nurse coders, blinded to study arm, will code parent-reported discharge diagnosis as (2) Correct, (1) Vague/Incomplete, or (0) Wrong/not concordant, by comparing it to diagnosis abstracted from discharge summary, using standard of whether a follow-up provider would know the diagnosis based on the parent-provided information; dichotomized for analysis.
Perceived Stress Scale | 2-6 weeks after discharge
  Scale score 0-16, using Perceived Stress Scale-Short Form 4-item measure; higher score indicates greater global stress and lower perceived control over it
Observed Communication: utterances in which team offers information | Day 1-5 of hospital admission
  Coding of audio-recorded communication with the medical team (on family centered rounds or similar discussion), reporting number of times in the discussion that a member of the medical team made an utterance that exchanged information with the family.
Observed Communication: utterances in which team offers supportive talk | Day 1-5 of hospital admission
  Coding of audio-recorded communication with the medical team (on family centered rounds or similar discussion), reporting number of times in the discussion that a member of the medical team made an utterance that was directly supportive of family
Observed Communication: utterances in which parent asks questions | Day 1-5 of hospital admission
  Coding of audio-recorded communication with the medical team (on family centered rounds or similar discussion), reporting number of times in the discussion that a parent or caregiver asks a question
Observed Communication: utterances in which parent responds assertively | Day 1-5 of hospital admission
  Coding of audio-recorded communication with the medical team (on family centered rounds or similar discussion), reporting number of times in the discussion that a parent or caregiver responds to something a member of the medical team says in an assertive manner
Observed Communication: parent talk-time | Day 1-5 of hospital admission
  Coding of audio-recorded communication with the medical team (on family centered rounds or similar discussion), reporting the percent of the overall discussion time during which the parent or caregiver was speaking
Observed Communication: global partnership rating | Day 1-5 of hospital admission
  Likert scale rating from 1-5 of audio-recorded communication with the medical team (on family centered rounds or similar discussion), rating the overall degree of partnership between family and medical team demonstrated during the discussion
30-day readmissions | 30 days after discharge from index hospital stay
  Readmissions to observation or inpatient status at the same hospital within 30 days of discharge from the index hospital stay

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Seattle Children's, Seattle, Washington